CLINICAL TRIAL: NCT00060710
Title: Phase II Study of CP-461 in the Treatment of Patients With Advanced Melanoma
Brief Title: CP-461 in the Treatment of Patients With Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Cell Pathways (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-461-013
Record Dates: First submitted 2003-05-09; First posted 2003-05-13 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Malignant Melanoma
Keywords: melanoma
MeSH Terms: conditions — Melanoma | interventions — (5-fluoro-2-methyl-1-(4-pyridyl)methylene-3-(N-benzyl)-indene)-acetamide hydrochloride

INTERVENTIONS:
Drug: CP-461

SUMMARY:
The purpose of this study is to determine the efficacy of CP-461 given twice daily orally in patients with advanced or metastatic malignant melanoma and to evaluate the safety profile of CP-461 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant melanoma that is advanced or metastatic.
* Patients may have received up to 2 prior systemic chemotherapy regimens (including dacarbazine, and alternative dosing schedule of temozolomide). The last chemotherapy must have been at least 4 weeks prior to study drug administration.
* Prior radiation therapy will be allowed. Radiotherapy must have been completed at least 4 weeks prior to study drug administration.
* Patients may have received prior surgery. At least 4 weeks must have elapsed and patients must have recovered from all side effects associated with surgery.
* Patients with measurable disease. At least one bidimensionally measurable lesion with clearly defined margins documented by: medical photograph for skin and oral lesions, plain X-ray with at least one diameter 0.5 cm or greater, CT, MRI, or palpation with both diameters 2 cm or greater. A radiated bony lesion may not be considered an evaluable lesion, unless there is evidence of disease progression at that site prior to administration of study drug.
* Clinical parameters: Life expectancy > 2 months, Age >18 years, ECOG performance status 0-2
* Patients should have adequate organ function related to the following: White count > 3000/ul, Platelet count > 70,000/ul, Hemoglobin > 8 g/l, Bilirubin WNL, AST and ALT < 2.5 x ULN, and Creatinine < 1.5 x ULN or 24 hour creatinine clearance > 60 ml/min
* There should be no acute infection requiring systemic antibiotics.
* Informed consent: Each patient must be completely aware of the nature of his/her disease process and must willingly give consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts.

Exclusion Criteria:

* Subjects who have brain metastases.
* More than 2 prior chemotherapy regimens for the treatment of advanced melanoma.
* Chemotherapy within four weeks prior to study drug administration.
* Radiation therapy to greater than or equal to 50% of the bone marrow. Patients must not have had prior radiotherapy to areas of measurable disease unless they have clearly progressive disease in this site or there is measurable disease outside the area of prior radiation.
* Insufficient recovery from all active toxicities of prior therapies.
* Subjects who are poor medical risks because of active nonmalignant systemic disease.
* Frequent vomiting or medical condition that could interfere with oral medication intake (e.g. partial bowel obstruction).
* No prior malignancy other than curatively treated carcinoma in-situ of the cervix or skin cancer. If in the opinion of the treating physician, sufficient time has elapsed, such that it is extremely likely that the patient has been cured of a prior malignancy, the patient may be eligible for the protocol.
* No serious medical or psychiatric illness preventing informed consent or intensive treatment (e.g. serious infection). HIV status or other severe illnesses will be assessed using medical records.
* Pregnant or nursing women. Both women and men must take adequate precautions to prevent pregnancy during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2003-01; Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia Presbyterian Medical Center, New York, New York, United States